CLINICAL TRIAL: NCT02148666
Title: Labelling of Stem Cells With Technetium 99- m Hexamethylene Propylene Amine Oxide ( Tc99m HMPAO)to Monitor Homing in the Human Heart. Bench to Bedside Studies [ COLT -- COronary Labelling Trial ]
Brief Title: Study of Homing of Labelled Stem Cells in Human Heart.
Acronym: COLT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: All India Institute of Medical Sciences (Other)
Collaborators: Indian Council of Medical Research (Other Government)
Responsible Party: Principal Investigator, Dr Sandeep Seth, Professor, All India Institute of Medical Sciences
Other Study IDs: ICMR 80/1/2014- BMS
Record Dates: First submitted 2014-05-23; First posted 2014-05-28 (Estimated); Last update posted 2014-06-09 (Estimated); Status verified 2014-06

CONDITIONS: Homing of Stem Cells in the Infarct Area.

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- experimental : intracoronary stem cells: intracoronary stem cells will be injected in infarct related artery.

SUMMARY:
One of the challenges of stem cell therapy is to understand the fate of the injected stem cell. By labelling various stem cells with radioisotopes their fate (homing) can be demonstrated. In this study, we will develop and refine the existing techniques of stem cell labelling to various subtypes of stem cells namely- freshly aspirated bone marrow cells, cryopreserved bone marrow cells, g-csf mobilized peripheral blood stem cells and umbilical cord cells. After testing the labelling efficacy and viability, these cells will be injected in to the coronary arteries of patients with myocardial infarction who have undergone a successful revascularization either by angioplasty or thrombolysis. Homing of stem cells will be demonstrated by nuclear scan after the procedure. We are adapting techniques used to label cells for detection of infection and bleeding using nuclear scans for in vivo scanning. Also we are using Technetium instead of FDG which has very little radioactivity allowing us to work with the current cardiac labs with out having to reconstruct the labs with special shielding for radioactive compounds. Real benefit of stem cells then can be explored after demonstrating the proper homing.

DETAILED DESCRIPTION:
Phase One: Four Different types of stem cells will be tested ( Freshly aspirated Bone marrow cells, cryopreserved cells, umbilical cord cells, Stem cells mobilised from bone marrow by g-csf, mesenchymal cells), and the efficacy of labelling documented and effect on viability noted. 3 samples of each type will be tested and the results will be documented. Different cells are being tried to test the efficiency of the labelling technique in different types of cells. This will provide the protocols for all future labelling studies. This will be conducted in collaboration between the stem cell department, nuclear medicine department and nuclear cardiology department.

Phase Two (Clinical Study):

This will be the pilot clinical study done alongside with the phase one study, and will enrol 10 patients with Recent Myocardial infarction ( within 3 months) . A small fraction of patient's own bone marrow stem cells will be labelled with Technetium 99m HMPAO. The labelled cells will be administered via the intracoronary injection along with the unlabeled stem cells. The localization of the radio-labelled stem cells in the myocardium will then be detected using the conventional Gamma camera.

ELIGIBILITY:
Inclusion Criteria:

* Myocardial Infarction (< Three Months) with either angioplasty or thrombolysis done to open the infarct causing artery.
* Patent coronary arteries after the infarct
* Left ventricular dysfunction (ejection fraction < 50%)

Exclusion Criteria:

* Ongoing infection
* Obstructive coronary disease
* History of symptoms more than 3 months
* Any evidence of malignancy or other systemic illness.
* Cell yield less than 10 million cells

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients within 3 months following myocardial infarction
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2014-08; Primary Completion 2017-08 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
homing of labelled cells to infarct zone and scan showing radioactivity in the infarct area | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Sandeep Seth, DM, Principal Investigator — All India Institute of Medical Sciences; Neeraj Parakh, DM, Study Chair — All India Institute of Medical Sciences; Chetan Patel, Study Chair — All India Institute of Medical Sciences; Sujata Mohanty, Study Chair — All India Institute of Medical Sciences; Sneh Lata, Study Chair — All India Institute of Medical Sciences; Balram Bhargava, DM, Study Chair — All India Institute of Medical Sciences; Vinay Kr Bahl, DM, Study Chair — All India Institute of Medical Sciences; Balram Airan, DM, Study Chair — All India Institute of Medical Sciences
Locations (1):
- All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Background] Huikuri HV, Kervinen K, Niemela M, Ylitalo K, Saily M, Koistinen P, Savolainen ER, Ukkonen H, Pietila M, Airaksinen JK, Knuuti J, Makikallio TH; FINCELL Investigators. Effects of intracoronary injection of mononuclear bone marrow cells on left ventricular function, arrhythmia risk profile, and restenosis after thrombolytic therapy of acute myocardial infarction. Eur Heart J. 2008 Nov;29(22):2723-32. doi: 10.1093/eurheartj/ehn436. Epub 2008 Oct 9. PMID 18845667
- [Background] Kraitchman DL, Tatsumi M, Gilson WD, Ishimori T, Kedziorek D, Walczak P, Segars WP, Chen HH, Fritzges D, Izbudak I, Young RG, Marcelino M, Pittenger MF, Solaiyappan M, Boston RC, Tsui BM, Wahl RL, Bulte JW. Dynamic imaging of allogeneic mesenchymal stem cells trafficking to myocardial infarction. Circulation. 2005 Sep 6;112(10):1451-61. doi: 10.1161/CIRCULATIONAHA.105.537480. Epub 2005 Aug 29. PMID 16129797
- [Background] Kang WJ, Kang HJ, Kim HS, Chung JK, Lee MC, Lee DS. Tissue distribution of 18F-FDG-labeled peripheral hematopoietic stem cells after intracoronary administration in patients with myocardial infarction. J Nucl Med. 2006 Aug;47(8):1295-301. PMID 16883008